CLINICAL TRIAL: NCT03472742
Title: An Observational Follow-Up Study of Patients Previously Enrolled in ADR-001-01 Study Against Liver Cirrhosis
Brief Title: An Follow-Up Study of Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Rohto Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ADR-001-02
Record Dates: First submitted 2018-03-01; First posted 2018-03-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-07

CONDITIONS: Decompensated Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Mesenchymal Stem Cell — As this is a follow-up and an observation study, ADR-001 was administered in the previous study, not in this study.
  Other Names: ADR-001

SUMMARY:
This is a follow-up study to assess safety and preliminary clinical activity of ADR-001 in patients with liver cirrhosis (Child-Pugh score; Grade B) caused by Hepatitis C or Nonalcoholic Steatohepatitis. Patients who have already participated in the ADR-001-01 study and completed the last evaluation after 24 weeks of administration will be eligible to this study.

Patients registered will continue follow-up observation and evaluate long-term safety and exploratory efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis patients enrolled in ADR-001-01 study and completed the last observation of the study
* Voluntary signed informed consent

Exclusion Criteria:

* Patients evaluated by investigators as inappropriate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Decompensated Liver Cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs) and serious AEs (SAEs) | Change from Baseline (Day 0) until 80 weeks
  An AE is any untoward medical event for the patient in the clinical study, associated with study medication. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of hospitalization, results in disability/incapacity, congenital anomaly/birth defect will be evaluated as an SAE.

SECONDARY OUTCOMES:
Change of liver function evaluated by Child-Pugh Score | Day 0, 28 weeks and 80 weeks (optional 12 weeks and 54 weeks)
  Change of liver function from the baseline will be evaluated by Child-Pugh score.
Improvement rate of Child-Pugh score | Day 0, 28 weeks and 80 weeks (optional 12 weeks and 54 weeks)
  Improvement rate of Child-Pugh score from the baseline will be evaluated.
Improvement rate of Child-Pugh grade | Day 0, 28 weeks and 80 weeks (optional 12 weeks and 54 weeks)
  Improvement rate of Child-Pugh grade from the baseline will be evaluated.
Number of patients with abnormal systolic blood pressure (SBP) and diastolic blood pressure (DBP) findings | Day 0, 28 weeks and 80 weeks (optional 12 weeks and 54 weeks)
  SBP and DBP will be measured at specific time points (mmHg)
Number of patients with abnormal pulse rate findings | Day 0, 28 weeks and 80 weeks (optional 12 weeks and 54 weeks)
  Pulse rate will be measured at specific time points (bit per minutes).
Number of patients with abnormal body temperature findings | Day 0, 28 weeks and 80 weeks (optional 12 weeks and 54 weeks)
  Axillary temperature will be measured at specific time points. (degree Celsius)
Number of patients with abnormal electrocardiogram (ECG) findings | Day 0, 28 weeks and 80 weeks (optional 12 weeks and 54 weeks)
  12-lead ECG will be obtained at specific time points.
Number of patients with abnormal clinical chemistry parameters | Day 0, 28 weeks and 80 weeks (optional 12 weeks and 54 weeks)
  Laboratory assessment for clinical chemistry parameters will include blood total protein, albumin, total and direct bilirubin, aspartate aminotransferase, alanine aminotransferase, r-glutamyltranspeptidase, alkaline phosphatase, cholinesterase, lactate dehydrogenase, uric acid, blood urea nitrogen, ammonia, serum creatinine, sodium, potassium, chlorine, calcium, phosphate, magnesium, C reactive protein creatinine, glucose,
Number of patients with abnormal clinical hematology parameters | Day 0, 28 weeks and 80 weeks (optional 12 weeks and 54 weeks)
  Laboratory assessment for clinical hematology will include white blood cell, red blood cell, hemoglobin, hematocrit, platelet, reticulocytes, neutrophils, lymphocytes, eosinophils, basophils, monocytes
Number of patients with abnormal urinalysis parameters | Day 0, 28 weeks and 80 weeks (optional 12 weeks and 54 weeks)
  Laboratory assessment for urinalysis will include glucose, protein and occult blood

CONTACTS AND LOCATIONS:
Locations (1):
- Niigata University Medical & Dental Hospital, Niigata, Japan